CLINICAL TRIAL: NCT03889665
Title: Influencia Del Entrenamiento en suspensión en el Equilibrio de Adultos jóvenes Sanos
Brief Title: Effects of Suspension Training on the Balance of Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Jose María Blasco Igual, Principal Investigator, University of Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRX-Balance
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspension training group (Experimental)
  Interventions: Other: Suspension training

INTERVENTIONS:
Other: Suspension training — Nine sessions of suspension training The suspension device will be TRX (R) The intervention will be administered in work:rest intervals (2:1) A global training approach will seek to train lower limbs, upper body and core musculature

SUMMARY:
Non-specific training through the use of devices in which the subject can be suspended is a technique that has aroused a growing interest in recent years. One of its advantages may be to enhance the balance, since it induces a high level of neuromuscular stimulation. Indeed, a suspension training suppose a high demand of the core musculature, require a high degree of postural control, precise response strategies , anticipatory capacity and muscular conditioning. However, current literature targeting healthy young adults and appraising the specifics effects of suspension training on balance is scarce or non-existent to the best of our knowledge. For this reason this interventional study will primarily assess the effects of suspension training on different balance components.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults aged between 18 and 30

Exclusion Criteria:

* Professional athlete
* Musculoskeletal injury in the last 6 months (i.e. sprain, bone fracture)
* Known balance disorders including vertigo, central or vestibular limitations

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Y-Balance test | Change from baseline to four weeks
  Measure of dynamic balance

SECONDARY OUTCOMES:
Emery test | Change from baseline to four weeks
  A timed test for static-dynamic balance assessment, the participant stands on one leg over a foam with closed eyes
Posturography measures | Change from baseline to four weeks
  Using a T-Plate pedometer
Jumping sideways test | Change from baseline to four weeks
  A measure to assess motor coordination under time pressure

OTHER OUTCOMES:
Five times sit-to-stand test | Change from baseline to four weeks
  This is generally used to assess the functional strength of the lower extremities, the transition movements, the balance and the risk of falls are evaluated
Stabilizer pressure biofeedback | Change from baseline to four weeks
  This is used to assess core strength

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat de València, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided